CLINICAL TRIAL: NCT03146936
Title: Swiss Primary Sclerosing Cholangitis Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Fondazione Epatocentro Ticino (Other)
Responsible Party: Sponsor
Other Study IDs: SASL40 - Swiss PSC Cohort
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Cholangitis, Sclerosing; PSC; Primary Sclerosing Cholangitis (PSC)
Keywords: PSC; Primary Sclerosing Cholangitis; Cohort
MeSH Terms: conditions — Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — 1. Serum (BD Vacutainer® SST II Advance)
  2. RNA (PAXgene™ Blood RNA tube- 762165)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Research project in which biological material is sampled and health-related personal data is further used and collected.

Coded data are used.

DETAILED DESCRIPTION:
The investigators wish to collect high quality prospective data on a rare disease in order to elucidate epidemiology, natural history, response to treatment and outcome. In addition, a biobank allows addressing specific scientific issues on a variety of open questions. The cohort will provide a platform for carrying out scientific research projects on PSC. In addition, the cohort will allow collaborations with reference networks on PSC abroad

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PSC according to established criteria (European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases) of any age. Patients not fulfilling such criteria but still diagnosed with PSC in a hepatology referral centre can be included
* patients living in Switzerland

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: PSC patients living in Switzerland of any age Patients diagnosed with PSC according to established criteria (European Association for the Study of the Liver. EASL Clinical Practice Guidelines: management of cholestatic liver diseases). Only patients living in Switzerland are enrolled. Enrollment of minors is possible upon consent of legal guardian
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-02-28 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease course | 3 years
  Observing disease course
Disease features | 3 years
  Observing disease features in Swiss population and see if they are similar to other countries'
Response to treatment | 3 years
  Observing response to treatment
Overall survival | 3 years
  Observing overall survival
Transplantation-free survival rate | 3 years
  Observing transplantation-free survival rate

CONTACTS AND LOCATIONS:
Locations (21):
- Switzerland (21):
  - Fondazione Epatocentro Ticino, Lugano, Canton Ticino
  - Gastroenterologie und Hepatologie Clarunis - Universitäres Bauchzentrum Universitätsspital Basel, Basel
  - Universitäts-Kinderspital beider Basel UKBB, Gastroenterologie&Ernährung, Basel
  - Inselspital, Bern
  - Kinderklinik, INSELSpital, Universität Bern, Pädiatrische Gastroenterologie, Hepatologie und Ernährung, Bern
  - Spital Bülach, Bülach
  - Kantonsspital Graubünden, Chur
  - Hôpitaux Universitaires de Genève, Centre Suisse des Maladies du foie de l'Enfant- Département de l'Enfant et de l'Adolescent, Geneva
  - Hôpitaux Universitaires de Genève, Service de Gastroentérologie & Hépatologie, Département des Spécialités, Geneva
  - CHUV: Centre hospitalier universitaire vaudois, Lausanne
  - CHUV Département femme-mère-enfant, Lausanne
  - Kantonsspital Baselland, Liestal
  - Kinderspital Luzern LUKS, Pädiatrische Gastroenterologie, Lucerne
  - Luzerner Kantonsspital, Lucerne
  - EOC Ospedale Regionale di Lugano - Italiano, Lugano
  - Ostschweizer Kinderspital, Sankt Gallen
  - Kantonsspital St.Gallen, Sankt Gallen
  - Kantonsspital Winterthur, Winterthur
  - Pädiatrische Gastroenterologie Departement Kinder- und Jugendmedizin Kantonsspital Winterthur, Winterthur
  - Universitäts-Kinderspital Zürich - Eleonorenstiftung, Zurich
  - Universitätsspital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No